CLINICAL TRIAL: NCT04238546
Title: Major Adverse Limb Events in Patients With Femoro-popliteal and Below-the-knee Peripheral Arterial Disease Treated With Either Sirolimus-coated Balloon or Standard Uncoated Balloon Angioplasty
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nils Kucher (Other)
Responsible Party: Sponsor-Investigator, Nils Kucher, Prof. Dr. med., University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SirPAD Trial
Record Dates: First submitted 2020-01-15; First posted 2020-01-23 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sirolimus-coated group (Experimental)
  Interventions: Device: sirolimus-coated balloon catheter
- Uncoated group (Active Comparator)
  Interventions: Device: uncoated balloon catheter

INTERVENTIONS:
Device: sirolimus-coated balloon catheter — angioplasty with sirolimus-coated balloon catheter
  Arms: Sirolimus-coated group
Device: uncoated balloon catheter — angioplasty with uncoated balloon catheter
  Arms: Uncoated group

SUMMARY:
The SirPAD trial is an academic, investigator-initiated, single-center, randomized, non-inferiority, open-label clinical trial investigating whether the use of sirolimus-coated balloon catheters in patients with peripheral artery disease of the femoro-popliteal or below-the-knee segment is not inferior to that of uncoated balloon catheters for major clinical outcomes (unplanned major amputation, target limb re-vascularization) and may provide advantages concerning important secondary outcomes, which will be evaluated using a pre-specified hierarchical order as part of the primary analysis.

DETAILED DESCRIPTION:
Peripheral artery disease (PAD) is a progressive atherosclerotic disease with symptoms ranging from intermittent claudication (IC) to critical limb ischemia (CLI). The majority of symptomatic PAD patients present with atherosclerotic lesions located in the femoro-popliteal arteries and endovascular therapy is the primary choice if the stenosis/occlusions involve <25 cm of the vessel. A minority of symptomatic PAD patients would present with infra-popliteal (distal or below-the-knee) lesions: in these patients, the endovascular treatment is challenging.

Drug-coated balloons (DCB) and drug-eluting stents (DES) were developed to prevent neo-intimal proliferation and restenosis after percutaneous transluminal angioplasty (PTA), an objective which had been achieved by the local application of either cytostatic (e.g. paclitaxel - a cytoskeletal disruptor) or immunosuppressive (e.g. sirolimus/everolimus - both mTOR inhibitors) substances on the vessel wall.

Over the past decade, a few randomized controlled trials (RCT) compared the efficacy and safety of drug-coated (mainly paclitaxel-coated) devices vs. that of uncoated ones, and demonstrated a significant reduction in restenosis rates, late lumen loss, and incidence of target lesion re-vascularization. However, the size of these trials was often too small to draw firm conclusions concerning major clinical outcomes. Moreover, substantial heterogeneity of the study populations and too restrictive eligibility criteria limited their external validity, leading to a difficult interpretation of the results of later meta-analyses. Indeed, these trials adopted as the primary outcome surrogate (and rather subjective) outcomes, such as vessel patency and target limb re-vascularization, which may be difficult to objectively adjudicate in the setting of an open-label trial, rather than ´hard´ objective clinical endpoints, such as major amputation or urgent revascularization due to critical limb ischemia.

Moreover, despite the short-term effects appeared promising based on imaging outcome, tthe results of a recent meta-analysis of 28 trials showed an increased two-year mortality in the group of patients treated with paclitaxel-coated balloons. Based on these results, and after analysis of follow-up data from the trials that led to the approval of these products, a Food and Drug Administration (FDA) panel concluded that, despite the short-term benefits with paclitaxel-based devices, safety concerns may exist for mid-term mortality risk.

Alternative drug candidates to paclitaxel-coated balloon catheters are the so-called limus-based analogs, which own cytostatic properties and are characterized by a wider therapeutic window. Recently, a novel balloon catheter has been CE-certified: it encapsulates sirolimus in phospholipid drug nanocarriers to improve adhesion properties of sirolimus and to provide better bioavailability. Similarly to paclitaxel-coated and uncoated devices, sirolimus-coated devices are currently approved for routine use in PAD and reimbursed in Switzerland.

The aim of the present trial is to compare the efficacy, as defined by a composite of clinically relevant non-subjective ´hard´ outcomes (major amputation and target lesion re-vascularization for critical limb ischemia), of sirolimus-coated vs. uncoated balloon angioplasty for peripheral artery disease in patients scheduled for infra-inguinal re-vascularization and selected based on a very limited number of inclusion criteria (all comers) aiming at maximization of external validity.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patients requiring endovascular angioplasty for PAD located below the inguinal ligament
* Written informed consent obtained from participant or legal guardian prior to randomization; in patients requiring emergency interventional treatment who are temporarily not capable of providing informed consent, consent will be subsequently obtained after the procedure if strict conditions apply. These include the assessment of the presumed will and patient decree, and requires the allocation of an independent physician

Exclusion Criteria:

* Pregnancy, breastfeeding, or planned pregnancy within the trial period or women of childbearing potential not using an adequate method of contraception
* Patients with known intolerance or allergy to sirolimus
* Participation in this or other clinical trials during the previous 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2020-11-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
unplanned major amputation of the target limb | one year
  An unplanned major amputation is defined as any amputation above the ankle on the target limb, which was not planned or not expectable at the time of screening or randomization. Patients with scheduled amputation undergoing re-vascularization to improve wound healing are referred to as planned amputation and will not count for the primary outcome
endovascular or surgical target lesion re-vascularization for critical limb ischemia | one year
  Critical limb ischemia is defined according to a Fontaine stage (classes III-IV)

SECONDARY OUTCOMES:
composite of unplanned (major or minor) index-limb amputations or any target lesion re-vascularization within 365 days after enrolment | one year
  Unplanned major amputation is defined analogously to the definition used for the primary efficacy endpoint

OTHER OUTCOMES:
Death from all causes | up to five years
  Death from all causes within 30 days, 180 days, one year, two years, and five years
Serious adverse events (SAEs) | one year
  Serious adverse events (SAEs) during initial hospitalization, within 180 days, and within 365 days
Serious adverse device related events (SADE) | up to one month
  Serious adverse device related events (SADE) during initial hospitalization
A composite of all-cause death and MALE | one month
  A composite of all-cause death and MALE within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Nils Kucher, Prof., Principal Investigator — University of Zurich
Locations (2):
- Switzerland (2):
  - University hospital zurich, Zurich, Canton of Zurich
  - HFR Fribourg - Hôpital Cantonal / Kantonsspital, Fribourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barco S, Sebastian T, Voci D, Engelberger RP, Grigorean A, Holy E, Leeger C, Munger M, Periard D, Probst E, Spescha R, Held U, Kucher N. Major adverse limb events in patients with femoro-popliteal and below-the-knee peripheral arterial disease treated with either sirolimus-coated balloon or standard uncoated balloon angioplasty: a structured protocol summary of the "SirPAD" randomized controlled trial. Trials. 2022 Apr 21;23(1):334. doi: 10.1186/s13063-022-06242-8. PMID 35449070